CLINICAL TRIAL: NCT06527456
Title: Intervention With General Practitioners to Improve Women's Participation in Cervical Cancer Screening
Acronym: INDIGO
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Intercommunal Creteil (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: INDIGO
Record Dates: First submitted 2023-10-20; First posted 2024-07-30 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: Cervical Cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- usual practice (No Intervention): the doctor will use their usual practices to encourage screening.
- Intervention (Experimental): the general practitioner or one of the professionals on their team will contact the patient (phone call, SMS, email, etc.), to encourage them to make an appointment to carry out the screening
  Interventions: Other: participation of the general practitioner

INTERVENTIONS:
Other: participation of the general practitioner — participation of the general practitioner in encouraging cervical cancer screening
  Arms: Intervention

SUMMARY:
In France, cervical cancer is the 12th most common female cancer with nearly 3,000 new cases per year.

Since 2018, a national Organized Cervical Cancer Screening program (DOCCU) has been set up and concerns all asymptomatic women aged 25 to 65.

This program, managed by the Regional Cancer Screening Coordination Centers (CRCDC), invites women who have not taken a sample within the recommended time frame to consult for screening. However, only 59% of patients participated.

The intervention of the general practitioner, an essential player in prevention, could allow for better awareness.

The objective of the INDIGO study is to evaluate the effectiveness of the intervention of a general practitioner on the participation rate in the DOCCU of patients who are not up to date with their screening.

DETAILED DESCRIPTION:
This is a cluster-randomized trial. Randomization will be performed at the GP practice level to limit the potential contamination bias between doctors within the same practice. GP practices will be randomized either to the 'usual practice' arm or the 'intervention' arm."

If they are in the "intervention" group, they or one of the professionals in their team will contact the patient (phone call, SMS, email, etc.), to encourage her to make an appointment to carry out the screening. Contact arrangements are left to the discretion of each general practitioner..

If they are in the "Usual practice" group, they will use their usual practices to encourage screening.

ELIGIBILITY:
Inclusion Criteria:

* Woman aged 25 to 65 living in Ile-De-France
* Eligible for DOCCU (not hysterectomized, not followed for a pre-cancerous or cancerous lesion of the cervix)
* Having declared the investigating general practitioner as a treating physician (MT) and whose MT practices in the territory of a CPTS in the UPEC area
* Affiliate to a social security scheme or beneficiary of such a scheme

Exclusion Criteria:

* Patient already included in a study on DOCCU
* Patient excluded from organized screening (cervical cancer, hysterectomy).
* Patient's opposition to participating in the study

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11200 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
screening participation rate | 12 month
  percentage of patients who had a screening Cervical Sample (cytology or HPV test within a timeframe satisfying the HAS recommendations according to age) among patients eligible for screening aged 25 to 65 years